CLINICAL TRIAL: NCT00390793
Title: Phase II Study of Combination of Hyper-CVAD and Dasatinib in Patients With Philadelphia (Ph) Chromosome Positive and/or BCR-ABL Positive Acute Lymphoblastic Leukemia (ALL)
Brief Title: Combination Chemotherapy and Dasatinib in Treating Participants With Philadelphia Positive or BCR-ABL Positive Acute Lymphoblastic Leukemia.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0478; NCI-2018-01846 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2006-0478 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2006-10-18; First posted 2006-10-20 (Estimated); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Acute Lymphoblastic Leukemia; BCR-ABL1 Fusion Protein Expression; Blast Phase Chronic Myelogenous Leukemia, BCR-ABL1 Positive; Philadelphia Chromosome Positive; Recurrent Acute Lymphoblastic Leukemia; t(9;22)
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Blast Crisis | interventions — Cyclophosphamide; Cytarabine; Dasatinib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Methotrexate; merphos; Prednisone; deltacortene; prednylidene; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (chemotherapy, dasatinib) (Experimental): See detailed description in outline.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dasatinib; Drug: Dexamethasone; Drug: Doxorubicin; Drug: Methotrexate; Drug: Prednisone; Drug: Vincristine

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Drug: Cytarabine — Given IV or IT
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Drug: Dexamethasone — Given IV or PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
Drug: Doxorubicin — Given IV
  Other Names: Adriablastin; Hydroxyl Daunorubicin; Hydroxyldaunorubicin
Drug: Methotrexate — Given IV or IT
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
Drug: Prednisone — Given PO
  Other Names: .delta.1-Cortisone; 1, 2-Dehydrocortisone; Adasone; Cortancyl; Dacortin; DeCortin; Decortisyl; Decorton; Delta 1-Cortisone; Delta-Dome; Deltacortene; Deltacortisone; Deltadehydrocortisone; Deltasone; Deltison; Deltra; Econosone; Lisacort; Meprosona-F; Metacortandracin; Meticorten; Ofisolona; Orasone; Panafcort; Panasol-S; Paracort; PRED; Predicor; Predicorten; Prednicen-M; Prednicort; Prednidib; Prednilonga; Predniment; Prednisonum; Prednitone; Promifen; Servisone; SK-Prednisone
Drug: Vincristine — Given IV
  Other Names: LEUROCRISTINE; VCR; Vincrystine

SUMMARY:
This phase II trial studies how well combination chemotherapy and dasatinib works in treating participants with Philadelphia-positive or B-cell receptor-ABL positive acute lymphoblastic leukemia. Drugs used in chemotherapy, such as cyclophosphamide, vincristine, doxorubicin, dexamethasone, methotrexate, and cytarabine, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Dasatinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving chemotherapy in combination with dasatinib may work better in treating participants with Philadelphia-positive or BCR-ABL positive acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the clinical efficacy (event-free survival) of an intensive short-term chemotherapy regimen (Hyper- cyclophosphamide, vincristine, doxorubicin, dexamethasone [CVAD] program) given in combination with the tyrosine kinase inhibitor dasatinib for Philadelphia (Ph)-positive and/or B-cell receptor BCR-ABL-positive acute lymphoblastic leukemia (ALL).

II. To evaluate other clinical efficacy (overall response rate and survival) and safety of an intensive short-term chemotherapy regimen (Hyper-CVAD program) given in combination with the tyrosine kinase inhibitor dasatinib for Philadelphia (Ph)-positive and/or BCR-ABL-positive acute lymphoblastic leukemia (ALL).

OUTLINE:

HYPER-CVAD THERAPY: Participants receive cyclophosphamide intravenously (IV) twice daily (BID) over 3 hours on days 1-3, vincristine IV over 30 minutes on days 4 and 11, and doxorubicin IV over 24-48 hours on day 4. Participants also receive dexamethasone orally (PO) or IV over 30 minutes on days 1-4 and 11-14, and dasatinib PO once daily (QD) on days 1-14 of course 1 and on days 1-21 for subsequent courses. Courses repeat every 21 days for up to 4 odd courses (1, 3, 5, and 7) in the absence of disease progression or unacceptable toxicity.

METHOTREXATE PLUS CYTARABINE: Participants receive methotrexate IV over 24 hours on day 1, dasatinib PO on days 1-21, and cytarabine IV BID over 2 hours on days 2 and 3. Courses repeat every 21 days for up to 4 even courses (2, 4, 6, and 8) in the absence of disease progression or unacceptable toxicity.

MAINTENANCE THERAPY: Participants receive vincristine IV over 30 minutes on day 1, prednisone PO on days 1-5, and dasatinib PO BID. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. During courses 6 and 13, participants may receive an additional course of hyper-CVAD therapy.

After completion of study treatment, participants are followed for up to 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of one of the following: Previously untreated Ph-positive acute lymphoblastic leukemia (ALL) (either t(9;22) and/or BCR-ABL positive) (includes patients initiated on first course of hyper-CVAD before cytogenetics known). These groups will be analyzed separately. After 1-2 courses of chemotherapy with or without imatinib mesylate (Gleevec). If they achieved complete response (CR), they are assessable only for event-free and overall survival, or if they failed to achieve CR, they are assessable for CR, event-free, and overall survival. Patients with relapsed Ph-positive ALL or lymphoid blast phase of chronic myelogenous leukemia (CML)
* Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* Adequate liver function (bilirubin less than or equal to 3.0 mg/dl, unless considered due to tumor), and renal function (creatinine less than or equal to 3.0 mg/dl, unless considered due to tumor)
* Adequate cardiac function as assessed clinically
* Signed informed consent

Exclusion Criteria:

* Active serious infection not controlled by oral or intravenous antibiotics
* Treatment with any investigational antileukemic agents or chemotherapy agents in the last 7 days before study entry, unless full recovery from side effects has occurred or patient has rapidly progressive disease judged to be life-threatening by the investigator
* Active secondary malignancy other than skin cancer (e.g., basal cell carcinoma or squamous cell carcinoma) that in the investigator's opinion will shorten survival to less than 1 year
* Active grade III-V cardiac failure as defined by the New York Heart Association criteria. Uncontrolled angina, or myocardial infarction (MI) within 6 months. Diagnosed or suspected congenital long QT syndrome. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes). Prolonged corrected QT (QTc) interval on pre-entry electrocardiogram (> 470 msec). Patients currently taking drugs that are generally accepted to have a risk of causing Torsades de Pointes (unless these can be changed to acceptable alternatives)
* Prior history of treatment with dasatinib
* Pregnant and lactating women will not be eligible; women of childbearing potential should have a negative pregnancy test prior to entering on the study and be willing to practice methods of contraception. Women do not have childbearing potential if they have had a hysterectomy or are postmenopausal without menses for 12 months. In addition, men enrolled on this study should understand the risks to any sexual partner of childbearing potential and should practice an effective method of birth control
* History of significant bleeding disorder unrelated to cancer, including:

  * Diagnosed congenital bleeding disorders (e.g., von Willebrand's disease)
  * Diagnosed acquired bleeding disorder within one year (e.g., acquired anti-factor VIII antibodies)
* Patients with documented significant pleural or pericardial effusions unless they are thought to be secondary to their leukemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2006-09-28 (Actual); Primary Completion 2024-02-02 (Actual); Study Completion 2024-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farhad Ravandi-Kashani, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Ravandi F, O'Brien S, Thomas D, Faderl S, Jones D, Garris R, Dara S, Jorgensen J, Kebriaei P, Champlin R, Borthakur G, Burger J, Ferrajoli A, Garcia-Manero G, Wierda W, Cortes J, Kantarjian H. First report of phase 2 study of dasatinib with hyper-CVAD for the frontline treatment of patients with Philadelphia chromosome-positive (Ph+) acute lymphoblastic leukemia. Blood. 2010 Sep 23;116(12):2070-7. doi: 10.1182/blood-2009-12-261586. Epub 2010 May 13. PMID 20466853
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Chemotherapy, Dasatinib)
Started | 107
Completed | 107
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy, Dasatinib)
Number analyzed (Participants) | 107
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 87
  >=65 years | 20
Age, Continuous [Median (Full Range); unit: years] | 53 [21 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 60
  More than one race | 0
  Unknown or Not Reported | 30
Region of Enrollment [Number; unit: participants]
  United States | 107

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival Rate (EFS)
Description: Time from date of treatment start until the date of failure or death from any cause.
Time Frame: Up to 17 years, 4 months, 2 days
Population: Of the 107 participants registered on study, 106 were evaluable for Event Free Survival.
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Chemotherapy, Dasatinib)
Number analyzed (Participants) | 106
Months | 21.3 [0.2 to 208]

2. Primary Outcome: Disease-free Survival
Description: Time from date of treatment start until the date of first objective documentation of disease-relapse.
Time Frame: Up to 17 years, 4 months, 2 days
Population: Of the 107 participants registered on study, 95 were evaluable for Disease Free Survival.
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Chemotherapy, Dasatinib)
Number analyzed (Participants) | 95
Months | 25.3 [0.3 to 208]

3. Secondary Outcome: Participants With a Response
Description: Participants achieving complete remission (CR) + partial remission (PR) - Complete Remission (CR): Normalization of the peripheral blood and bone marrow with 5% or less blasts in normocellular or hypercellular marrow with a granulocyte count of 1 x 10^9/L or above, and platelet count of 100 x 10^9/L. Complete resolution of all sites of extramedullary disease is required for CR.
Time Frame: Up to 17 years, 4 months, 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy, Dasatinib)
Number analyzed (Participants) | 106
Participants | 95

4. Secondary Outcome: Overall Survival
Description: Time from date of treatment start until date of death due to any cause or last Follow-up.
Time Frame: Up to 17 years, 4 months, 2 days
Population: Of the 107 participants registered on study, 106 were evaluable for Overall Survival.
Measure: Median (Full Range); unit: Months
Arm/Group | Treatment (Chemotherapy, Dasatinib)
Number analyzed (Participants) | 106
Months | 42.9 [0.2 to 208]

ADVERSE EVENTS:
Time Frame: Up to 17 years, 4 months, 2 days
Arm/Group | Treatment (Chemotherapy, Dasatinib)
All-Cause Mortality (participants affected / at risk) | 4/107
Serious Adverse Events (participants affected / at risk) | 38/107
Other Adverse Events (participants affected / at risk) | 0/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Chemotherapy, Dasatinib) (N=107)
abdominal Pain (Gastrointestinal disorders) | 2 (2)
Bilateral Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cellulitis buttocks (Infections and infestations) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (2)
Death (General disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Diverticulitis (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Entercoccal Bacteremia (Infections and infestations) | 1 (1)
Facial Pain (General disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 8 (10)
Fracture Ribs (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 3 (3)
Hematemesis (Gastrointestinal disorders) | 1 (1)
Hematothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (3)
Infection (Infections and infestations) | 2 (3)
Jaw Pain (General disorders) | 1 (1)
Miocardial Infarction (Cardiac disorders) | 1 (1)
Mucositis (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Nausea/Vomiting (Gastrointestinal disorders) | 4 (4)
Neutropenic Fever (Blood and lymphatic system disorders) | 13 (18)
Pain (General disorders) | 1 (1)
Perianal Pain (Gastrointestinal disorders) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Pneumonia (Infections and infestations) | 5 (6)
Positive West Niles Virus (General disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Septic Shock (Infections and infestations) | 2 (3)
Shoulder/Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Subdural Hematoma (Vascular disorders) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 3 (3)
Weakness (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2009-06-23): https://cdn.clinicaltrials.gov/large-docs/93/NCT00390793/Prot_SAP_000.pdf